CLINICAL TRIAL: NCT03988608
Title: A Non-randomized, Open-label, Multi-center, Phase II Study to Assess the Safety and Efficacy of Eltrombopag in Chinese Subjects With Refractory or Relapsed Severe Aplastic Anemia
Brief Title: Study Assessed the Safety and Efficacy of Eltrombopag in Chinese Refractory or Relapsed Severe Aplastic Anemia (SAA) Subjects.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CETB115E2202
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-01

CONDITIONS: Aplastic Anemia
Keywords: Severe Aplastic Anemia; Eltrombopag; ETB115; Chinese subject; Chinese refractory or relapsed SAA subjects; refractory severe aplastic anemia; relapsed severe aplastic anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eltrombopag (Experimental): Subjects started eltrombopag treatment at 25 mg/day since Day 1.
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag are film-coated tablets containing 25 mg of eltrombopag free acid in each tablet.
  Other Names: ETB115

SUMMARY:
This was a non-randomized, open-label, phase II study to assess the efficacy and safety of eltrombopag in Chinese subjects with refractory or relapsed severe aplastic anemia (SAA). Treatment with eltrombopag was started at 25 mg/day and increased by 25 mg/day every 2 weeks according to the platelet count up to 150 mg/day. The hematological response rate was assessed at 3, 6 months and 1 year after starting the study treatment (Week 13, 26 and 52).

DETAILED DESCRIPTION:
This was a bridging study to support China registration. An estimation strategy rather than a formal hypothesis testing was pursued. Twenty subjects were enrolled into the study.

Treatment with eltrombopag started at 25 mg/day and increased by 25 mg/day every 2 weeks according to the platelet count, up to 150 mg/day. Hematological response rate was assessed at 3, 6 months and 1 year (Week 13, 26 and 52) after starting the study treatment. Subjects in whom the treatment was found to be effective at 6 months continued to receive the treatment. Eltrombopag was discontinued if the treatment was ineffective at 6 months. Subjects discontinued eltrombopag before 6 months if any of the treatment discontinuation criteria was met.

Analysis set for the primary endpoint was Full Analysis Set (FAS) and subjects who discontinue from the study before Week 26 were treated as non-responders in the response analysis. Eltrombopag treatment was provided to subjects who were considered to require continued treatment at Week 26. After Week 26, if all of the hematologic response criteria (i.e., platelet count > 50×109/L, hemoglobin level > 100 g/L without transfusion, and neutrophil count > 1.0×109/L) remained fulfilled for more than 8 weeks, the dose of eltrombopag was decreased by half. If the response continued for further 8 weeks even at the decreased dose, the treatment was discontinued. If a decrease in any of the hematologic values (i.e., platelet count < 30×109/L, hemoglobin < 90 g/L, or neutrophil count < 0.5×109/L) was found after dose reduction, the dose was increased to the previous level. Furthermore, after treatment interruption, the treatment was restarted if any of the hematologic values decreased to the above-mentioned levels. The response assessment and safety evaluation were performed at Week 52.

The Extension part of this study started 1 year (Week 52) after the initiation of study treatment. This part was included in the study with an ethical consideration for subjects who required continued treatment. The continued treatment was provided up to the launch of eltrombopag after approval. Follow-up visit was performed 30 days after the discontinuation of eltrombopag treatment.

To better understand the pharmacokinetics (PK) characteristics of eltrombopag in Chinese severe aplastic anemia (SAA) patient population, intensive PK blood samples were collected only in the initial 12 Chinese subjects receiving 25 mg/day dose after reaching steady-state, to provide evaluable full PK profiles. Steady-state trough concentrations were collected at other dose levels and in other subjects.

ELIGIBILITY:
Inclusion Criteria:

* Chinese patients aged greater than or equal to 18 years old.
* Patient with a previous diagnosis of severe aplastic anemia and had insufficient response following at least one treatment course in the period time of > 6 months of immunosuppression with a regimen containing anti-thymocyte globulin (ATG), anti-lymphocyte globulin (ALG), and/or cyclophosphamide, or alemtuzumab.
* Platelet count ≤ 30 × 10^9/L at screening.
* Patient must not currently have the option of stem cell transplantation.
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Patient with QTcF (Fridericia's QT correction formula) at screening <450 msec, or <480 msec with bundle branch block, as determined via the mean of a triplicate ECG and assessed at site.

Exclusion Criteria:

* Treatment with ATG/ALG, cyclophosphamide or alemtuzumab in the past 6 months.
* Congenital aplastic anemia
* AST or ALT ≥3 times the upper limit of normal.
* Creatinine, total bilirubin, and alkaline phosphatase (ALP) ≥ 1.5× local ULN (total bilirubin ≥ 2.5 × local ULN with Gilbert's Syndrome).
* Paroxysmal nocturnal hemoglobinuria (PNH) granulocyte clone size determined by flow cytometry ≥ 50%.
* Presence of chromosomal aberration (-7/7q- detected by fluorescence in situ hybridization (FISH), or other aberrations detected by G-band staining).
* Evidence of a clonal hematologic bone marrow disorder on cytogenetics.
* Past medical history of thromboembolism within 6 months or current use of anticoagulants.
* Have any concomitant malignancies and must be fully recovered from treatment for any other malignancy and have been disease-free for 5 years.
* Patient with clinically significant (of such severity that it would preclude the patient's ability to consent, be compliant with study procedures, tolerate protocol therapy) bacterial, fungal, mycobacterial, parasitic or viral infection (Patient with acute bacterial infections requiring antibiotic use should delay Screening/enrollment until the course of antibiotic therapy has been completed).
* Patient with known hepatocellular disease
* Presences of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening.
* Cardiac disorder (NYHA) functional classification Grade II/III/IV
* Past medical history of immediate or delayed hypersensitivity to compounds chemically similar to eltrombopag or their excipients.
* Treatment with another investigational product within 30 days.
* Prior treatment with eltrombopag, romiplostim, or any other TPO (thrombopoietin) receptor agonist.
* Positive result for HIV (Human Immunodeficiency Virus) antibody test.
* Pregnant or nursing (lactating) woman.
* Woman of child-bearing potential.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2023-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- China (4):
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Tianjin

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Chang H, He G, Fu R, Li F, Han B, Li T, Liu L, Mittal H, Jin H, Zhang F. Efficacy and safety of eltrombopag in Chinese patients with refractory or relapsed severe aplastic anemia. Sci Rep. 2023 Nov 2;13(1):18955. doi: 10.1038/s41598-023-45607-0. PMID 37919313
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2080

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled all 20 participants from 5 sites in China.
Pre-assignment Details: One of the main criteria for enrollment was for Chinese patients aged ≥ 18 years, previously diagnosed with SAA and who had insufficient response following at least one treatment course in the period time of > 6 months of immunosuppression with a regimen containing anti-thymocyte globulin (ATG), anti-lymphocyte Immunoglobulin (ALG), and/or cyclophosphamide, or alemtuzumab.
Groups:
- Eltrombopag: Participants started eltrombopag treatment at 25 mg/day from Day 1 and increased by 25 mg/day every 2 weeks according to the platelet count up to 150 mg/day.
Period: Overall Study
Arm/Group | Eltrombopag
Started | 20
Completed 26-week Treatment Phase | 17
Entered Week 52 Treatment Phase | 15
Completed Week 52 Treatment Phase | 14
Completed | 14
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 3
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) comprised all patients to whom study treatment had been assigned and received one dose of study treatment.
Arm/Group | Eltrombopag
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (13.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 20

OUTCOME MEASURES:

1. Primary Outcome: Hematologic Response Rate at 6 Months (Week 26) by Investigator
Description: Hematologic response rate: percentage of subjects who met any of the International Working Group criteria: Platelet count: If platelet transfusion independent at baseline (BL): Transfusion independent and increase from BL by 20×10^9/L or more; If platelet transfusion dependent at BL: No platelet transfusion requirement for 8 weeks; Hemoglobin: If red blood cells (RBC) transfusion independent at BL: transfusion independent and increase from BL by 15 g/L or more; If RBC transfusion dependent at BL: A decrease of at least 4 units in RBC transfusions in the post-treatment 8-week period (1 unit = RBC derived from 200 mL blood) or no RBC transfusion requirement for 8 weeks; Neutrophil count: In the absence of granulocyte colony stimulating factor (G-CSF) taken within 21 days preceding the blood sample collection: Increase from BL by 0.5×10^9/L or more, or (if < 0.5×10^9/L at BL) increase by 100% or more. Patients who discontinued from the trial before week 26 were treated as non-responders.
Time Frame: 6 months (Week 26)
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment had been assigned and received one dose of study treatment. The patients who discontinued from the trial before Week 26 were treated as non-responders.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 20
Percentage of participants | 70.0 [49.2 to 86.0]

2. Secondary Outcome: Hematologic Response Rate by Investigator
Description: Hematologic response rate: percentage of subjects who met any of the International Working Group criteria: Platelet count: If platelet transfusion independent at baseline (BL): Transfusion independent and increase from BL by 20×10^9/L or more; If platelet transfusion dependent at BL: No platelet transfusion requirement for 8 wks; Hemoglobin: If red blood cells (RBC) transfusion independent at BL: transfusion independent and increase from BL by 15 g/L or more; If RBC transfusion dependent at BL: A decrease of at least 4 units in RBC transfusions in the post-treatment 8-week period (1 unit =RBC derived from 200 mL blood) or no RBC transfusion requirement for 8 wks; Neutrophil count: In the absence of granulocyte colony stimulating factor (G-CSF) taken within 21 days preceding the blood sample collection: Increase from BL by 0.5×10^9/L or more, or (if < 0.5×10^9/L at BL) increase by 100% or more. Patients who discontinued from the trial before wks 13 & 26 were treated as non-responders.
Time Frame: Week (Wk) 13, Week 52
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment had been assigned and received one dose of study treatment.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 20
Percentage of participants
  Week 13 | 65.0 [44.2 to 82.3]
  Week 52 | 65.0 [44.2 to 82.3]

3. Secondary Outcome: Change From Baseline in Platelet Count
Description: Change (increase from baseline) in platelet count (in the absence of platelet transfusion) were calculated according to the lab test results entered into the case report form (CRF) that were summarized at each visit using descriptive statistics. Platelet Count (×109/L) was assessed in hematology test.
Time Frame: Baseline, Week 13, Week 26, Week 52
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment had been assigned and received one dose of study treatment.
  These were the patients in FAS with a valid assessment for the outcome measure at baseline and at Weeks 13, 26 and 52.
Measure: Mean (Standard Deviation); unit: 10^9 platelets/liter
Arm/Group | Eltrombopag
Number analyzed (Participants) | 20
10^9 platelets/liter
  Baseline (BL) | 10.725 (7.8731)
  Change from BL at Week 13/Day92: number analyzed (Participants) | 17
  Change from BL at Week 13/Day92 | 10.265 (14.1456)
  Change from BL at Week 26/Day 183: number analyzed (Participants) | 15
  Change from BL at Week 26/Day 183 | 26.933 (30.5304)
  Change from BL at Week 52/Day 365: number analyzed (Participants) | 14
  Change from BL at Week 52/Day 365 | 41.071 (56.6816)

4. Secondary Outcome: Change From Baseline in Hemoglobin Levels
Description: Change (increase from baseline) in hemoglobin (in the absence of red blood cell (RBC) transfusion) were calculated according to the lab test results entered into the CRF that were summarized at each visit using descriptive statistics. Hemoglobin level (g/L) was assessed in hematology test.
Time Frame: Baseline, Week 13, Week 26 and Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: gram/liter
Arm/Group | Eltrombopag
Number analyzed (Participants) | 20
gram/liter
  Baseline | 66.9 (19.90)
  Change from BL at Week 13/Day92: number analyzed (Participants) | 14
  Change from BL at Week 13/Day92 | 22.4 (23.47)
  Change from baseline at Week 26/Day 183: number analyzed (Participants) | 13
  Change from baseline at Week 26/Day 183 | 31.9 (29.20)
  Change from BL at Week 52/Day 365: number analyzed (Participants) | 14
  Change from BL at Week 52/Day 365 | 32.9 (33.21)

5. Secondary Outcome: Change From Baseline in Neutrophil Count
Description: Change (increase from baseline) in neutrophil count (in the absence of granulocyte colony stimulating factor (G-CSF) and calculated according to the lab test results entered into the CRF that were summarized at each visit using descriptive statistics). Neutrophil count (×109/L) was assessed in hematology test.
Time Frame: Baseline, Week 13, Week 26 and Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 10^9 neutrophils/liter
Arm/Group | Eltrombopag
Number analyzed (Participants) | 20
10^9 neutrophils/liter
  Baseline | 1.199 (1.3483)
  Change from BL at Week 13/Day 92 (n = 16): number analyzed (Participants) | 16
  Change from BL at Week 13/Day 92 (n = 16) | -0.160 (1.4141)
  Change from baseline at Week 26/Day 183 (n = 14): number analyzed (Participants) | 14
  Change from baseline at Week 26/Day 183 (n = 14) | 0.196 (1.6822)
  Change from BL at Week 52/Day 365 (n = 14): number analyzed (Participants) | 14
  Change from BL at Week 52/Day 365 (n = 14) | 0.447 (1.5764)

6. Secondary Outcome: Time to Hematologic Response by Investigator
Description: Time to hematological response was defined as the time from the date of first study drug administration to the first hematological response.
  If a participant did not meet hematological response before or at the cutoff date, censoring was performed using the date of last assessment.
Time Frame: Baseline to Week 26
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment had been assigned and received one dose of study treatment and achieved a hematologic response.
Measure: Median (90% Confidence Interval); unit: Weeks
Arm/Group | Eltrombopag
Number analyzed (Participants) | 20
Weeks | 10.0 [8.0 to 12.0]

7. Secondary Outcome: Duration of Hematologic Response by Investigator
Description: Duration of hematologic response (any response according to the response criteria for the primary endpoint). For subjects who responded, duration of response was defined as the number of weeks from the first date of hematological response until the first date of relapse or death. Only participants with at least two response assessments were included for the duration of hematologic response assessment.
Time Frame: up to approx. 3.5 years
Population: Participants in the FAS who achieved a hematologic response. The Full Analysis Set (FAS) comprised all patients to whom study treatment had been assigned and received one dose of study treatment and achieved a hematologic response.
Measure: Median (90% Confidence Interval); unit: Weeks
Arm/Group | Eltrombopag
Number analyzed (Participants) | 15
Weeks | NA [22.3 to NA] — NA: Not estimable due to insufficient number of participants with events

8. Secondary Outcome: Frequency of Platelets Transfusion
Description: For subjects receiving transfusion (platelets) at baseline, the frequency of platelet transfusion in each period (Baseline: 4 weeks before Day 1; Week 13, 26, 52: 4 weeks before each visit day) was summarized using descriptive statistics.
Time Frame: Baseline, Week 13, Week 26 and Week 52
Population: Participants in the FAS who were platelet transfusion dependent at baseline and who did not discontinue prior to the corresponding visit date (Week 13, 26 and 52).
Measure: Mean (Standard Deviation); unit: occurrences
Arm/Group | Eltrombopag
Number analyzed (Participants) | 10
occurrences
  Baseline | 1.8 (1.32)
  Week 13: number analyzed (Participants) | 9
  Week 13 | 0.4 (0.88)
  Week 26: number analyzed (Participants) | 8
  Week 26 | 0.1 (0.35)
  Week 52: number analyzed (Participants) | 6
  Week 52 | 0.0 (0.00)

9. Secondary Outcome: Amount of Platelets Transfusion
Description: The amount of transfusion was defined as the sum of transfusion multiplied by the volume of transfusion.
Time Frame: Baseline, Week 13, Week 26 and Week 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Eltrombopag
Number analyzed (Participants) | 10
Units
  Baseline | 3.7 (3.63)
  Week 13: number analyzed (Participants) | 9
  Week 13 | 0.4 (0.88)
  Week 26: number analyzed (Participants) | 8
  Week 26 | 0.1 (0.35)
  Week 52: number analyzed (Participants) | 6
  Week 52 | 0.0 (0.00)

10. Secondary Outcome: Frequency of Red Blood Cells (RBC) Transfusion
Description: For subjects receiving transfusion (RBC (Red Blood Cell)) at baseline, the frequency of RBC transfusion in each period (Baseline: 8 weeks before Day 1; Week 13, 26, 52: 8 weeks before each visit day) was summarized using descriptive statistics.
Time Frame: Baseline, Week 13, Week 26 and Week 52
Population: Participants in the FAS who were RBC transfusion dependent at baseline and who did not discontinue prior to the corresponding visit date (Week 13, 26 and 52).
Measure: Mean (Standard Deviation); unit: occurrences
Arm/Group | Eltrombopag
Number analyzed (Participants) | 14
occurrences
  Baseline | 3.0 (2.04)
  Week 13: number analyzed (Participants) | 12
  Week 13 | 1.8 (2.83)
  Week 26: number analyzed (Participants) | 11
  Week 26 | 1.5 (2.02)
  Week 52: number analyzed (Participants) | 10
  Week 52 | 0.5 (0.71)

11. Secondary Outcome: Amount of Red Blood Cells (RBC) Transfusion
Description: The amount of RBC transfusion was defined as the sum of transfusion multiplied by the volume of transfusion.
Time Frame: Baseline, Week 13, Week 26 and Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Eltrombopag
Number analyzed (Participants) | 14
Units
  Baseline | 6.6 (4.16)
  Week 13: number analyzed (Participants) | 12
  Week 13 | 3.8 (6.18)
  Week 25: number analyzed (Participants) | 11
  Week 25 | 3.0 (4.02)
  Week 52: number analyzed (Participants) | 10
  Week 52 | 1.4 (1.90)

12. Secondary Outcome: Plasma PK Parameters of Eltrombopag: Cmax
Description: Cmax is the maximum (peak) observed plasma drug concentration after single dose administration (mass*volume-1). Blood samples were collected from patients to assess the plasma concentrations of eltrombopag. The plasma concentrations were used to determine the PK characteristics of eltrombopag. Serial intensive PK blood samples were collected for the initial 25 mg/day dose to provide at least 12 participants with evaluable PK profiles at steady state.
Time Frame: pre-dose, and 1, 2, 4, 6, 8 and 24 hours post-dose on Day 14
Population: Participants in the pharmacokinetic analysis set (PAS) who had an evaluable pharmacokinetic (PK) profile at steady state.
  The pharmacokinetic analysis set (PAS) included all patients who received at least one dose of eltrombopag and who had at least one evaluable PK sample.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Eltrombopag
Number analyzed (Participants) | 12
ng/mL | 3450 (1900)

13. Secondary Outcome: Plasma PK Parameters of Eltrombopag: Tmax
Description: Tmax is the time to reach maximum (peak) plasma drug concentration after single dose administration (time). Blood samples were collected from all patients to assess the plasma concentrations of eltrombopag. The plasma concentrations were used to determine the PK characteristics of eltrombopag. Serial intensive PK blood samples were collected for the initial 25 mg/day dose to provide at least 12 participants with evaluable PK profiles at steady state.
Time Frame: pre-dose, and 1, 2, 4, 6, 8 and 24 hours post-dose on Day 14
Population: as for outcome 12
Measure: Median (Full Range); unit: hour
Arm/Group | Eltrombopag
Number analyzed (Participants) | 12
hour | 3.73 [0.917 to 5.90]

14. Secondary Outcome: Plasma PK Parameters of Eltrombopag: AUCtau & AUClast
Description: AUCtau is the area under the curve calculated to the end of a dosing interval (tau) at steady-state (amount*time*volume-1). AUClast is the AUC calculated from time 0 to the time of the last quantifiable concentration. Blood samples were collected from patients to assess the plasma concentrations of eltrombopag. The plasma concentrations were used to determine the PK characteristics of eltrombopag. Serial intensive PK blood samples were collected for the initial 25 mg/day dose to provide at least 12 participants with evaluable PK profiles at steady state.
Time Frame: pre-dose, and 1, 2, 4, 6, 8 and 24 hours post-dose on Day 14
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Eltrombopag
Number analyzed (Participants) | 12
h*ng/mL
  AUCtau: number analyzed (Participants) | 11
  AUCtau | 67900 (31400)
  AUClast | 62700 (33200)

15. Secondary Outcome: Plasma PK Parameters of Eltrombopag: CLss/F
Description: Steady State (CLss/F) is the apparent systemic (or total body) clearance at steady state from plasma (volume/time) following drug administration. Blood samples were collected from patients to assess the plasma concentrations of eltrombopag. The plasma concentrations were used to determine the PK characteristics of eltrombopag. Serial intensive PK blood samples were collected for the initial 25 mg/day dose to provide at least 12 participants with evaluable PK profiles at steady state.
Time Frame: pre-dose, and 1, 2, 4, 6, 8 and 24 hours post-dose on Day 14
Population: Participants in the pharmacokinetic analysis set (PAS) who had an evaluable PK profile at steady state and who had a valid value for the outcome measure. The PAS included all patients who received at least one dose of eltrombopag and who had at least one evaluable PK sample.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Eltrombopag
Number analyzed (Participants) | 11
L/h | 0.441 (0.178)

16. Secondary Outcome: Plasma Trough Concentration of Eltrombopag
Description: Ctrough is the pre-dose concentration at the end of dose interval (mass*volume-1). Blood samples were collected from patients to assess the plasma concentrations of eltrombopag. The plasma concentrations were used to determine the PK characteristics of eltrombopag. Serial intensive PK blood samples were collected for the initial 25 mg/day dose to provide at least 12 participants with evaluable PK profiles at steady state. Sparse PK blood samples were collected for the other doses and in the rest of the patients for Ctrough assessment.
Time Frame: Pre-dose sample on the 15th day after each new dose level was started
Population: The pharmacokinetic analysis set (PAS) included all patients who received at least one dose of eltrombopag and who had at least one evaluable PK sample.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Eltrombopag
Number analyzed (Participants) | 20
ng/mL
  concentration at 25 mg | 2180 (1490)
  concentration at 50 mg: number analyzed (Participants) | 16
  concentration at 50 mg | 5180 (3320)
  concentration at 75 mg: number analyzed (Participants) | 19
  concentration at 75 mg | 11300 (6000)
  concentration at 100 mg: number analyzed (Participants) | 19
  concentration at 100 mg | 14700 (8070)
  concentration at 125 mg: number analyzed (Participants) | 15
  concentration at 125 mg | 20300 (11300)
  concentration at 150 mg: number analyzed (Participants) | 15
  concentration at 150 mg | 23800 (13700)

17. Secondary Outcome: Number of Participants With Clonal Evolution
Description: Number of participants with clonal evolution with a normal karyotype at baseline including clonal evolution to PNH (Paroxysmal Nocturnal Hemoglobinuria), evolution to AML (Acute Myeloid Leukemia) or MDS (Myelodysplastic Syndromes).
Time Frame: From Baseline up to approx. 2.9 years
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment had been assigned.
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 20
Participants | 2

18. Post Hoc Outcome: All Collected Deaths
Description: Deaths were collected from the first dose until end of study, a maximum duration of up to 3.5 years.
  On-treatment deaths were collected within 30 days of the last dose, while post-treatment deaths were collected more than 30 days after the last dose for those who discontinued treatment early.
  Adverse events were collected from the first dose until 30 days after the last dose, also up to a maximum duration if 3.5 years.
  Adverse Events were not collected in the post-treatment period.
Time Frame: On-treatment deaths: up to approx. 3.5 years, post-treatment deaths: up to approx. 3.5 years
Population: All enrolled participants.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 20
Participants
  All Deaths | 1
  On-treatment deaths | 0
  Post-treatment deaths | 1

ADVERSE EVENTS:
Time Frame: Deaths were collected from the first dose until end of study, a maximum duration of up to 3.5 years. On-treatment deaths were collected within 30 days of the last dose, while post-treatment deaths were collected more than 30 days after the last dose for those who discontinued treatment early. Adverse events were collected from the first dose until 30 days after the last dose, also up to a maximum duration if 3.5 years. Adverse Events were not collected in the post-treatment period.
Description: Any sign or symptom that occurs during the conduct of the trial and safety follow-up. Deaths in the post treatment survival follow-up are not considered Adverse Events.
Groups:
- Eltrombopag (On-treatment): Safety data collected from first dose of study medication up to 30 days after last dose.
- Eltrombopag (Post-treatment): Deaths collected from 31 days after last dose of study medication up to end of study. These are not considered adverse events.
Arm/Group | Eltrombopag (On-treatment) | Eltrombopag (Post-treatment)
All-Cause Mortality (participants affected / at risk) | 0/20 | 1/20
Serious Adverse Events (participants affected / at risk) | 8/20 | 0/0
Other Adverse Events (participants affected / at risk) | 19/20 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (On-treatment) (N=20) | Eltrombopag (Post-treatment) (N=0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | NA
Gastritis (Gastrointestinal disorders) | 1 | NA
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | NA
Pyrexia (General disorders) | 1 | NA
Liver injury (Hepatobiliary disorders) | 1 | NA
Pneumonia (Infections and infestations) | 3 | NA
Spermatic cord funiculitis (Infections and infestations) | 1 | NA
Upper respiratory tract infection (Infections and infestations) | 2 | NA
Intentional product misuse (Injury, poisoning and procedural complications) | 2 | NA
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | NA
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | NA
Syncope (Nervous system disorders) | 1 | NA
Abnormal uterine bleeding (Reproductive system and breast disorders) | 1 | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (On-treatment) (N=20) | Eltrombopag (Post-treatment) (N=0)
Cataract (Eye disorders) | 2 | NA
Diarrhoea (Gastrointestinal disorders) | 2 | NA
Mouth ulceration (Gastrointestinal disorders) | 2 | NA
Oedema peripheral (General disorders) | 3 | NA
Pyrexia (General disorders) | 5 | NA
Drug-induced liver injury (Hepatobiliary disorders) | 2 | NA
Hepatic function abnormal (Hepatobiliary disorders) | 4 | NA
Hyperbilirubinaemia (Hepatobiliary disorders) | 5 | NA
Liver injury (Hepatobiliary disorders) | 3 | NA
COVID-19 (Infections and infestations) | 3 | NA
Upper respiratory tract infection (Infections and infestations) | 8 | NA
Alanine aminotransferase increased (Investigations) | 3 | NA
Aspartate aminotransferase increased (Investigations) | 2 | NA
Blood bilirubin increased (Investigations) | 2 | NA
Blood creatinine increased (Investigations) | 6 | NA
Blood glucose increased (Investigations) | 4 | NA
Blood lactate dehydrogenase increased (Investigations) | 3 | NA
Electrocardiogram T wave abnormal (Investigations) | 2 | NA
Gamma-glutamyltransferase increased (Investigations) | 2 | NA
Glomerular filtration rate decreased (Investigations) | 2 | NA
Weight increased (Investigations) | 2 | NA
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | NA
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | NA
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4 | NA
Hyperuricaemia (Metabolism and nutrition disorders) | 5 | NA
Hyponatraemia (Metabolism and nutrition disorders) | 2 | NA
Hypoproteinaemia (Metabolism and nutrition disorders) | 2 | NA
Iron overload (Metabolism and nutrition disorders) | 2 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e., data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2019-09-02): https://cdn.clinicaltrials.gov/large-docs/08/NCT03988608/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-22): https://cdn.clinicaltrials.gov/large-docs/08/NCT03988608/SAP_001.pdf